CLINICAL TRIAL: NCT07272733
Title: Early Detection, Remote Augmented Reality Combined Rehabilitation Therapy, and Translational Therapy for Patients With Chronic Kidney Disease and Cognitive Disorder
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202208048; NSTC 112-2221-E-038-016 (Other Grant/Funding Number: Ministry of Science and Technology)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Disease (Stages 3b-5); Mild Cognitive Disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Neurocognitive Disorders | interventions — ketosteril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD stage 3-5 Age between 20-85 with mild cognitive disorder
  Interventions: Drug: Ketosteril

INTERVENTIONS:
Drug: Ketosteril — Ketosteril will lower protein binded uremic toxin

SUMMARY:
More than half of the patients with nephropathy have cognitive impairment, which can reach the level of dementia.The decline of renal function is more serious. With the aging of the population and changes in lifestyle, the number of patients is increasing day by day. The reasons are 1.Chronic kidney disease is prone to sarcopenia due to restricted protein intake, and even affects the heart and brain other than the kidneys. 2. Often accompanied by limb weakness and inconvenience of movement, sometimes it is very inconvenient to go to the hospital for treatment, so the hospital is the center cardio to perform telerehabilitation therapy is another option, so the purpose of this study is for patients with cognitive impairment Rehabilitation in virtual reality at a distance to evaluate its effectiveness. In this study, we selected from the treatment room of Beijing Medical Rehabilitation Department choose a space, simulate the situation of home telerehabilitation, and implement virtual reality telerehabilitation with the hospital as the center. The effect of distance rehabilitation and traditional rehabilitation. The study is expected to recruit 60 patients with chronic cognitive impairment and kidney disease who will be randomized. Divided into two groups A, B and C for training, 20 patients in each group, of which group A received ketoacid amino acid supplementation therapy, 3 capsules per day for 3 months; patients in group B received telerehabilitation for 30 minutes three days a week for a total of 3 months; C C The group was the control group, and the treatment was carried out according to the medical routine. The 60 patients received cognitive function,Brain functional MRI, balance ability, clinical function, clinical physical data, daily living function and depression Index evaluation. The results of this study can be used as a reference for future home tele-rehabilitation and ketoacid amino acid supplementation.

ELIGIBILITY:
Inclusion Criteria:

Chronic kidney disease stage 3-5

Exclusion Criteria:

* without cognitive disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
MMSE | Half a year
  Cognitive test

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No